CLINICAL TRIAL: NCT07281651
Title: Investigating the Role of Central Pain Hypersensitivity in Skeletal Muscle Neural Drive, in People With Knee Pain, and in People With Fibromyalgia Syndrome (Pain-Neural Drive)
Brief Title: Investigating the Role of Central Pain Hypersensitivity in Skeletal Muscle Neural Drive
Acronym: Pain-Drive
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Stephanie Smith, Dr Stephanie Smith, University of Nottingham
Other Study IDs: FMHS 36-1124 / FMHS 128-0425
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Knee Pain; Fibromyalgia
Keywords: Chronic Pain; Musculoskeletal Conditions; Fibromyalgia; Muscle Function; Physical Functioning; Disability; Central Aspects of Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Knee Pain: Adults with knee pain lasting over 3 months
  Interventions: Other: Central Pain Hypersensitivity
- Fibromyalgia: Adults with Fibromyalgia
  Interventions: Other: Central Pain Hypersensitivity
- Control Group: Adults without chronic pain conditions
  Interventions: Other: Central Pain Hypersensitivity

INTERVENTIONS:
Other: Central Pain Hypersensitivity — No intervention carried out

SUMMARY:
Background: pain lasting for 12 weeks or beyond, which is often referred to as chronic pain, is common for people living with musculoskeletal conditions (e.g. arthritis, low back pain and fibromyalgia). Pain is often not directly related to the degree of muscle or joint damage. Adaptations of the central nervous system (brain, spinal cord and nerves) often occur in chronic musculoskeletal conditions and can influence how we feel pain (central pain hypersensitivity). Pain can impact on muscle activity and movement. Muscle activity is also governed by nerve signals from the central nervous system (neural drive).

The goal of this cross-sectional observational study is to investigate whether chronic musculoskeletal pain is associated with altered nerve signalling (neural drive) to skeletal muscles in adults 40 years or over with chronic knee pain, fibromyalgia and healthy pain free volunteers.

The main questions it aims to answer are:-

* Is central pain hypersensitivity associated with altered nerve signalling to skeletal muscles in adults 40 years or over with chronic pain (knee pain and for fibromyalgia) as well as healthy volunteers?
* Is altered nerve signalling to skeletal muscles associated with physical function and disability?

Participants will be asked to:-

* Have sensory testing to determine how they feel pain
* Complete static leg and arm muscle contractions with electrodes on the skin to measure muscle electrical activity
* Complete questionnaires
* Perform a short set of mobility tasks including walking, rising from a chair and balancing.

DETAILED DESCRIPTION:
Participants will be required to attend two visits to Derby Medical School.

Screening and eligibility assessment:- Prior to booking an appointment to attend the study, potential participants will be given the opportunity to ask questions and be pre-screened for eligibility for the study.

Participation involves two study visits:- Visit 1 involves screening for eligibility, and providing informed consent. A brief history of pain condition and clinical knee assessment will be carried out. Familiarisation with the muscle testing protocol (practicing a set of muscle contractions) a questionnaire booklet will be provided at this visit. Visit 1 will last between 30 and 45 minutes.

Visit 2 is the test session. Body weight and height will be taken. Pain sensitivity testing (quantitative sensory testing) will be followed by neuromuscular testing while sitting in a specially designed chair. Isometric muscle contractions will be measured using an isometric dynamometer. One muscle will be tested in the lower legs and one muscle in the upper arms (on both sides).

Electrodes will be placed on a muscle at the front of the leg (tibialis anterior) and at the front of the upper arm (biceps brachii). A battery of isometric (static) muscle contractions will be performed following a force trace visual feedback on a monitor. To test whether experimental remote pain has an influence on neuromuscular functioning, a temporary pain stimulus will be applied to the arm via blood pressure cuff to a subjective level of 4/10 where '0' no pain and '10' worse pain or discomfort imaginable. A series of muscle contractions will be carried out during the remote discomfort stimulus lasting approximately 2 minutes. If discomfort becomes too much at any time the cuff will be removed immediately.

Physical performance and self-reported physical functioning and disability will be measured with a simple performance measure and questionnaires respectively. A pre-test questionnaire will be used to collect relevant data, including: pain severity, duration of pain condition, duration of pain, other medical conditions, gender, ethnicity, smoking status, employment status, use of pain medications. The questionnaire also includes validated questionnaires on quality of life, central aspects of pain, disability, physical functioning, fatigue and physical activity.

ELIGIBILITY:
Inclusion Criteria:

Knee pain group

* History of knee pain with an intensity level of 4 out of 10 or greater (where 0 is no pain and 10 is the worst pain imaginable) for most days in the past 3 months

Fibromyalgia group

* Fibromyalgia diagnosis (participant self-reporting a previous diagnosis by a clinician)
* Pain with an intensity level of 4 out of 10 or greater (where 0 is no pain and 10 is the worst pain imaginable) for most days in the past 3 months

Control group

- Pain free individuals without known osteoarthritis

Exclusion Criteria:

* BMI>35
* Body weight of 250kg or higher
* Pregnancy (women)
* Inability to give consent
* Inability to meet the requirements of clinical assessment
* Performed strenuous physical exercise in the past 24 hours prior to testing
* Consumed alcohol on day of testing
* Consumed caffeine on day of testing

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants may be recruited via various routes. Recruitment will primarily be through the Investigating Musculoskeletal Health and Wellbeing (IMH&W) cohort, which comprises over 7610 people with and without a range of musculoskeletal conditions. Participants with knee pain or fibromyalgia or healthy pain free individuals may be recruited via word of mouth, via University of Nottingham intranet and posters. Participant with fibromyalgia may be recruited to take part via local community support groups.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Once at baseline
  Pressure Pain Threshold as an index of central pain hypersensitivity.
  Pressure Pain Threshold (PPT) performed with digital algometer, applied at proximal forearm. A gradually increasing pressure is applied, and participants indicate when the sensation of pressure turns to pain. PPDT measured in Kilopascals (kPa). Three tests applied, which are then mean averaged. Lower PPT indicates greater pain sensitivity.
Temporal Summation | Once at baseline
  Temporal Summation as an index of central pain hypersensitivity.
  Temporal Summation (TS) assessed using a puncate stimulator (designed not to puncture the skin). Participants rate their experience of sharpness during the stimulus on a 10 cm visual analogue scale, first following one application, and second following 10 repeated applications. TS is calculated by subtracting first score from second (in cm). Higher positive scores indicate higher sensitivity.
Conditioned Pain Modulation | Once at baseline
  Conditioned Pain Modulation as an index of central pain hypersensitivity.
  Conditioned pain modulation (CPM) involves temporary ischaemic pain at one arm by way of blood pressure cuff. PPT simultaneously applied to opposite forearm. CPM calculated as conditioned PPT minus non-conditioned PPT in kilopascals (kPa). Lower positive or negative CPM indicates higher sensitivity.
Short Physical Performance Battery Test | Once at baseline
  A measure of physical performance of basic physical tasks, which is made up of for tasks:-
  Standing balance: participants are timed as to how long they can maintain standing balance unassisted without walking aids. First with feet side by side, second in semi-tandem stance, third in full tandem-stance. Points are awarded if balance is maintained for 10 seconds.
  Walking speed: participants are timed to walk a short distance (3 or 4 meters) at their usual walking pace. Allowed to use their usual walking aids. Points are awarded based on pre-set time scales for completing the walk.
  Repeated sit to stand: participants timed as to how many times they can sit to stand 5 times from an average height chair. Points awarded based on pre-set durations.
  Points are combined to give an overall score ranging from 0 - 12. A higher overall score = higher physical performance.
Motor Unit Firing Characteristics of skeletal muscles via High Density Surface Electromyography (HDsEMG) | Once at baseline
  Motor unit firing characteristics will be captured using HDsEMG during a range of sub-maximal skeletal muscle contractions. HDsEMG sensor will be placed on the skin over the muscles tibialis anterior and biceps brachii bilaterally to record muscle activation. Established methods will allow analysis of motor unit firing characteristics in terms of size, number, complexity, reliability and firing rate.

SECONDARY OUTCOMES:
Central Aspects of Pain Questionnaire | Once at baseline
  A self completed questionnaire giving a central aspects of pain factor, an index of central nervous system aspects of pain. The questionnaire includes 8 items covering neuropathic-like pain, fatigue, cognitive difficulty, catastrophizing, anxiety, sleep disturbance, depression and widespread pain. For the former 7 items, respondents rate the frequency of experiencing symptoms over the past week with four options "never", "sometimes", "often", "always". The widespread pain item involves shading areas of a manakin relating to painful areas of the body experienced on most days in the last four weeks. All items are combined to give an overall score. Scores can range from 0 to 16. The higher the score, the greater the central aspects of pain factor.
Neuromuscular control | Once at baseline
  A range of isometric muscle contraction patterns will be performed (tibialis anterior and biceps brachii) in terms of contraction strength, duration and rate of force generation. Neuromuscular control metrics will include force steadiness, and force accuracy.
Neuromuscular functioning alongside remote pain stimulus | Once at baseline
  To test whether experimental remote pain has an influence on neuromuscular functioning, a temporary pain stimulus will be applied to the arm via blood pressure cuff to a subjective level of 4/10 where '0' no pain and '10' worse pain or discomfort imaginable. A series of isometric (static) muscle contractions will be carried out during the remote discomfort stimulus lasting approximately 2 minutes. If discomfort becomes too much at any time the cuff will be removed immediately.
  The effect of remote pain stimulus on neuromuscular functioning will be analysed in terms of neuromuscular control (including force steadiness, and force accuracy) and motor unit firing characteristics (using HDsEMG).
Pain Intensity | Once via questionnaire prior to objective testing, however current pain level also completed on day of objective testing. Both are at baseline.
  Pain intensity measured by self-report using an 11 point numerical rating scale from 0-10, where 0 is no pain and 10 is the worst pain imaginable.
  Three items will be administered, using the 11 point scale detailed above:-
  * Over the past 4 weeks, how strong was your strongest pain?
  * Over the past 4 weeks, how strong was your pain on average?
  * How would you assess your pain now, at this moment?
RAND 36 Item Survey 1.0 - Physical Performance sub-scale (SF-36 PF) | Once at baseline.
  The RAND SF-36 PF is a sub-scale of the overall RAND SF-36 quality of life self-completed questionnaire. The SF-36 PF is a measure of Physical Functioning.
  There are 10 question covering a range of every day physical functioning activities. Three responses are possible regarding the level of limitation experienced for each item i.e. "not limited at all" (three points), "limited a little" (2 points) or "limited a lot" (1 point). The overall SF-36 PF score is from 0-100, where 100 indicates the most favourable health state.
Health Assessment Questionnaire - Disability Index (HAQ-DI) | Once at baseline
  The HAQ-DI is a self-completed questionnaire designed to measure a person's functional ability over the past week. It covers eight categories of daily activities, including:- Dressing and Grooming; Arising; Eating; Walking; Hygiene; Reach; Grip and Activities. It also asks questions on the use of aids or devices and the need for help from other people. Each item is scored from 0-3. The overall HAQ-DI score is calculated by summing all the domains, and dividing by eight, providing an ordinal score from 0 (no-disability) to 3 (severe disability).
Modified Fatigue Impact Scale (MFIS) | Once at baseline
  The MFIS is a self-completed questionnaire which provides a measure of how fatigue impacts on daily life. It has 21 items and provides an overall score out of 84 with higher scores indicating a greater impact of fatigue. Four sub-scales can be calculated: physical, cognitive and psychosocial, indicating how much fatigue impacts on these aspects of health and wellbeing.
Physical Activity Scale for the Elderly (PASE) | Once at baseline
  The PASE is a self-completed questionnaire which measures physical activity levels over the past 7 days. It includes activities relating to leisure, household and occupation. It provides an overall score from 0-400 or more and a higher score indicates higher levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Smith, PhD, Principal Investigator — University of Nottingham; Mathew Piasecki, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham Graduate Entry Medicine and Health, Royal Derby Hospital, Uttoxeter Road, Derby, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No